CLINICAL TRIAL: NCT01372501
Title: A Pilot Trial of Obese Subjects Previously Implanted With the EndoBarrier Gastrointestinal Liner
Brief Title: Study of Obese Subjects Previously Implanted With the EndoBarrier Gastrointestinal Liner
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-3
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: Device (Experimental): All patients will be implanted with the Endobarrier Liner device
  Interventions: Device: Endobarrier Liner

INTERVENTIONS:
Device: Endobarrier Liner — Medical device placed endoscopically in the duodenum
  Other Names: GI Sleeve

SUMMARY:
The purpose of this study is to determine whether the GI Endobarrier Liner can be reimplanted.

DETAILED DESCRIPTION:
Patients with obesity are at significantly greater risk of developing significant co-morbid complications, and are associated with an increased risk in all-cause mortality. The GI Endobarrier Liner represents a viable alternative to other short-term weight loss methods. It is a minimally invasive endoscopic procedure, which may allow patients to recover faster with less morbidity and mortality. This study is investigating whether the the GI Endobarrier Liner can be reimplanted.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 55 years - Male or Female
* Previously implanted with the EndoBarrier Gastrointestinal Liner
* Subjects willing to comply with trial requirements
* Subjects who have signed an informed consent form
* Women who are post-menopausal, surgically sterile or on oral contraceptives for the duration of the study and who do not plan on becoming pregnant during the course of the trial.

Exclusion Criteria:

* Treatment represents an unreasonable risk to the subject
* Pregnant or have intention of becoming pregnant for the duration of the trial
* Unresolved alcohol or drug addiction
* Subjects receiving weight loss medications (prescription, over-the- counter, or herbal dietary medications)
* Previous gastrointestinal surgery that could affect the ability to place the EndoBarrier Liner or the function of the implant.
* Subjects with active and uncontrolled gastroesophageal reflux disease (GERD)
* Subjects with symptomatic kidney stones prior to implant
* Subjects taking corticosteroids or drugs known to affect GI motility (i.e. Reglan)
* Subjects with iron deficiency and/or iron deficiency anemia
* History of Inflammatory bowel disease or condition of the gastrointestinal tract, such as ulcers or Crohn's disease
* Subjects with symptomatic gallstones prior to implant
* Symptomatic coronary artery disease or pulmonary dysfunction
* Known infection (Subjects who have a known infection at time of screening can be enrolled if the infection is treated prior to their procedure; if they still have an infection on day of procedure they must be withdrawn)
* History of congenital or acquired anomalies of the gastrointestinal tract such as atresias or stenoses
* Pancreatitis or other serious organic conditions
* Subjects requiring prescription anticoagulation therapy
* Subjects unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during the implant period
* Subject or Family history of a known diagnosis or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
* Participating in another ongoing investigational clinical trial
* Mentally retarded or emotionally unstable, or exhibits psychological characteristics requiring medication that affects appetite (i.e. tricyclic antidepressants and atypical antipsychotic medications) which, in the opinion of the Investigator, makes the subject a poor candidate for device placement or clinical trial.
* Subjects with active H. pylori (Note: Subjects may be enrolled if they had a prior history of H. Pylori and were successfully treated or are diagnosed during baseline tests and undergo successful treatment before their procedure)
* Subjects with or a history of coagulopathy, upper gastro-intestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex P Escalona, MD, Principal Investigator — Pontificia Universidad Catolica de Chile, Santiago, Chile
Locations (1):
- Dr. Alex P Escalona, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data is available on site at Sponsor

RESULTS

PARTICIPANT FLOW:
Groups:
- EndoBarrier Liner Device: All patients will be implanted with the Endobarrier Liner device.
  Endobarrier Liner: Medical device placed endoscopically in the duodenum
Period: Overall Study
Arm/Group | EndoBarrier Liner Device
Started | 19
Completed | 14
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Device migration | 1

BASELINE CHARACTERISTICS:
Groups:
- EndoBarrier Liner Device: All patients will be implanted with the Endobarrier Liner device
  Endobarrier Liner: Medical device placed endoscopically in the duodenum
Arm/Group | EndoBarrier Liner Device
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (11.32)
Gender [Count of Participants; unit: Participants]
  Female | 15
  Male | 4
Region of Enrollment [Number; unit: participants]
  Chile | 19

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the % Excess Weight Loss at Week 52 or Last Assessment
Description: Excess weight was determined from ideal body weights based on a BMI of 25 kg/m2
Time Frame: 52 Weeks
Population: Full Analysis Set (FAS) population had a device successfully implanted.
Measure: Mean (Standard Deviation); unit: %EWL
Arm/Group | EndoBarrier Liner Device
Number analyzed (Participants) | 19
%EWL | 26.9 (20.35)

2. Secondary Outcome: Change in Absolute Weight Loss From Baseline to Week 52
Time Frame: Week 52
Population: Per Protocol Population (n=14); subjects who had the device implanted for 52 weeks.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- EndoBarrier Liner Device: Endobarrier Liner: Medical device placed endoscopically in the duodenum
Arm/Group | EndoBarrier Liner Device
Number analyzed (Participants) | 14
kg | -7.1 (3.34)

ADVERSE EVENTS:
Time Frame: 1.5 years
Arm/Group | EndoBarrier Liner Device
Serious Adverse Events (participants affected / at risk) | 10/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier Liner Device (N=19)
Gastrointestinal infection (Gastrointestinal disorders) | 1 (1)
Upper abdominal pain (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier Liner Device (N=19)
Abdominal pain upper (Gastrointestinal disorders) | 11 (20)
Abdominal pain (Gastrointestinal disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 4 (4)
Pyrexia (General disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (4)
Gastroenteritis (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 10 (11)
Procedural vomiting (Injury, poisoning and procedural complications) | 8 (10)
Headache (Nervous system disorders) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No